CLINICAL TRIAL: NCT06094712
Title: An Open-Label, Single Dose Study to Evaluate the Pharmacokinetics of the Phase 2 Formulation of CORT125134 Capsules in Healthy Male Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of the CORT125134 Phase 2 Formulation in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CORT125134-122
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CORT125134 (Experimental): After an overnight fast, subjects will receive a single CORT125134 150-mg oral dose of the Phase 2 capsule formulation on Day 1.
  Interventions: Drug: CORT125134

INTERVENTIONS:
Drug: CORT125134 — CORT125134 150-mg capsule

SUMMARY:
A study designed to characterize the pharmacokinetic (PK) profile of CORT125134 following a single 150-mg oral dose of the Phase 2 capsule formulation of CORT125134 in 8 healthy male subjects.

DETAILED DESCRIPTION:
Following an overnight fast, subjects will be administered a single 150-mg oral dose of CORT125134 capsules on the morning of Day 1. Blood samples for determination of PK parameters will be collected predose and at serial time points up to 120 hours after study drug administration. The secondary objective of the study is to characterize the PK profile of metabolite CORT125201 following a single 150-mg oral dose of the Phase 2 capsule formulation of CORT125134 in 8 healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 kg/m^2 to 30 kg/m^2, inclusive, and body weight of ≥50 kg (110 pounds)
* Able to understand the study procedures, voluntarily consent to participate in this study, and provide written informed consent prior to start of any study-specific procedures
* Willing and able to remain in the study unit for the duration of the confinement period
* Must agree to use an adequate method of contraception as described in the protocol
* Must agree to study restrictions as defined in the protocol.

Exclusion Criteria:

* Subject and/or any of his immediate family members are employed by the study clinic, Corcept, or any subcontractor involved in this study
* Has a pregnant partner
* Has previously been enrolled in this study
* History of, and/or has been treated for, alcoholism, substance abuse, or drug abuse within the year prior to Day 1
* Positive screen for drugs of abuse or a positive alcohol result
* Current smokers and those who have smoked and/or used tobacco and/or nicotine containing products within the 6 months before Day 1 and are unable to refrain from using tobacco during the study treatment and evaluation period
* Clinically significant abnormality, in the Investigator's opinion, as indicated by the results of hematology, biochemistry, or urinalysis tests or from medical history, social history, vital signs, or physical examination
* Positive serology result for hepatitis B surface antigen (HbsAg), hepatitis C virus antibody (HCV Ab) or HIV
* Current or past history of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, gastrointestinal or neurological disease
* Active renal and/or hepatic disease
* Any form of cancer within the 2 years prior to study entry, with the exception of basal cell and/or squamous cell cancer of the skin that has been resected completely and is without evidence of local recurrence or metastasis
* History and/or symptoms of adrenal insufficiency
* History of jaundice and/or subject has had a cholecystectomy
* Active acute or chronic infectious diseases
* History of clinically significant gastrointestinal disease including gastroesophageal reflux disease, malabsorption syndrome, colon cancer, chronic colitis, Crohn's disease, inflammatory bowel disease, gastroparesis, constipation, chronic diarrhea, obstruction, gastrointestinal bleeding, and/or ulcers
* A condition such as asthma, chronic obstructive pulmonary disease, or a chronic inflammatory condition that could be aggravated by glucocorticoid (GC) blockade
* A QTcF interval of >450 msec (at Screening and/or Day -1)
* History of additional risk factors for torsade's de pointes (eg heart failure, hypokalemia, family history of long QT syndrome)
* Heart rate at rest of <45 bpm or >100 bpm (at Screening and/or Day -1)
* Sustained sitting systolic blood pressure >140 mmHg or <100 mmHg or a diastolic blood pressure >95 mmHg at Screening or Day -1
* Presence or history of clinically significant allergy that requires treatment; hay fever is allowed unless it is active
* Donation of blood or blood products (including plasma) during the 8 weeks before Day 1
* Has taken any prescribed and/or over-the-counter medication for which 5 times the medication's elimination half life will not be completed by Day 1, and/or herbal preparation in the 14 days before Study Day 1. Acetaminophen (up to 1 g per day) is permitted.
* Subjects who are taking a cytochrome P450 (CYP) 3A inducer (including herbal preparations such as St John's Wort), or have taken such treatment within 1 month before Day 1
* Are currently using GCs or have a history of GC use at any dose within the last 3 months or have a history of intraarticular GC within the last 6 months
* History or presence of any medical condition or disease which, in the opinion of the Investigator, could interfere with the conduct of the study or could put the subject at unacceptable risk
* Regular (daily) consumption of alcohol exceeding 2 bottles of beer or the equivalent amount of other forms of alcohol (1 serving = 12 oz beer, 5.0 oz wine, or 1.5 oz distilled spirits)
* Any use of alcohol within 48 hours of dosing on Day 1
* Use of any experimental or investigational drugs within 30 days prior to Day 1.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-04-27 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of plasma CORT125134 (Cmax) | Predose and at serial time points up to 120 hours after dosing
Time of maximum concentration of plasma CORT125134 (Tmax) | Predose and at serial time points up to 120 hours after dosing
Area under the concentration-time curve from time zero to the time of last measurable concentration of plasma CORT125134 (AUC0-last) | Predose and at serial time points up to 120 hours after dosing
Area under the concentration-time curve from time zero extrapolated to infinity of plasma CORT125134 (AUC0-inf) | Predose and at serial time points up to 120 hours after dosing
Apparent terminal half-life of plasma CORT125134 (T1/2) | Predose and at serial time points up to 120 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Hunt, Study Director — Corcept Therapeutics
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No